CLINICAL TRIAL: NCT02180061
Title: Phase Ib Study of MK-3475 in Subjects With Advanced Melanoma
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Advanced Melanoma (MK-3475-041/KEYNOTE-041)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-041; 142637 (Registry Identifier: JAPIC-CTI); MK-3475-041 (Other: Merck Protocol Number); KEYNOTE-041 (Other: Merck)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Melanoma
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advanced Cutaneous Melanoma (Experimental): Participants with advanced cutaneous melanoma received pembrolizumab, 2 mg/kg, intravenously (IV) over 30 minutes on Day 1 of each 3-week dosing cycle (Q3W).
  Interventions: Biological: Pembrolizumab
- Advanced Mucosal Melanoma (Experimental): Participants with advanced mucosal melanoma received pembrolizumab, 2 mg/kg, IV over 30 minutes on Day 1 Q3W.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475

SUMMARY:
This study will assess the safety, tolerability, and efficacy of every-3-week dosing (Q3W) of pembrolizumab (MK-3475) in participants with advanced melanoma; participants may receive pembrolizumab for up to 2 years if deriving clinical benefit. The primary study hypothesis is that treatment with single agent pembrolizumab will result in a clinically meaningful overall response rate.

DETAILED DESCRIPTION:
Participants who discontinue pembrolizumab after achieving a complete response (CR) and subsequently develop progressive disease (PD) may be eligible to enter a Second Course Phase and receive pembrolizumab again.

The end of the study for each participant will occur with: 1) the marketing approval of pembrolizumab for melanoma, 2) the completion of safety follow up or 3) the time when a possibility of entry to second course of treatment is lost, whichever occurs last.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of locally advanced (unresectable Stage III) or metastatic (Stage IV) melanoma not amenable to local therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least one measurable lesion
* Adequate organ function

Exclusion criteria:

* Prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-PD ligand-1 (PD-L1), anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) agent
* Is currently participating or has participated in a study with an investigational compound or device within 30 days, or 5X half-life of the investigational compound, whichever is longer, of initial dosing on this study
* Chemotherapy, targeted small molecule therapy, radiotherapy, or biological cancer therapy (including monoclonal antibodies) within 4 weeks prior to the first dose of trial treatment, or not recovered (<= Grade 1 or baseline) from adverse events due to a previously administered agent
* Expected to require any other form of systemic or localized antineoplastic therapy while in study
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
* Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 1 week prior to the first dose of study treatment
* Received a live vaccine within 4 weeks prior to the first dose of trial treatment
* Has a known hypersensitivity to the components of the study drug or another monoclonal antibody
* History or evidence of active pneumonitis
* Human immunodeficiency virus (HIV)-positive
* Has known history of active Hepatitis B or C
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial treatment through 120 days after the last dose of study medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yamazaki N, Takenouchi T, Fujimoto M, Ihn H, Uchi H, Inozume T, Kiyohara Y, Uhara H, Nakagawa K, Furukawa H, Wada H, Noguchi K, Shimamoto T, Yokota K. Phase 1b study of pembrolizumab (MK-3475; anti-PD-1 monoclonal antibody) in Japanese patients with advanced melanoma (KEYNOTE-041). Cancer Chemother Pharmacol. 2017 Apr;79(4):651-660. doi: 10.1007/s00280-016-3237-x. Epub 2017 Mar 11. PMID 28283736
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These results include data received prior to the safety database cutoff date of 23-Oct-2017.
Period: Overall Study
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
Started | 34 | 8
Completed | 9 | 0
Not Completed | 25 | 8
Not completed — Adverse Event | 4 | 2
Not completed — Clinical Progression | 5 | 1
Not completed — Progressive Disease | 15 | 5
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Advanced Cutaneous Melanoma: Participants with advanced cutaneous melanoma received pembrolizumab, 2 mg/kg, IV over 30 minutes on Day 1 Q3W.
- Total: Total of all reporting groups
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma | Total
Number analyzed (Participants) | 34 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (13.3) | 58.6 (15.5) | 63.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 21 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 8 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 8 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
Time Frame: All AEs: Up to 30 days after last dose of study drug; Serious AEs: Up to 90 days after last dose of study drug (Up to 27 months)
Population: The All Participants as Treated (APaT) population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
Number analyzed (Participants) | 34 | 8
Participants | 34 | 8

2. Primary Outcome: Number of Participants Discontinuing Treatment Due to AEs
Description: as for outcome 1
Time Frame: Up to last dose of study drug (Up to 24 months)
Population: The APaT population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
Number analyzed (Participants) | 34 | 8
Participants | 5 | 2

3. Primary Outcome: Overall Response Rate (ORR) Per Central Radiology Review Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: The ORR, using RECIST 1.1, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) at any time during the study, based on central radiology review.
Time Frame: Up to 24 months
Population: The Full Analysis Set (FAS) population consisted of all allocated participants who had measurable lesions at the Baseline scan as assessed by central radiology review and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
Number analyzed (Participants) | 29 | 8
Percentage of Participants | 24.1 [10.3 to 43.5] | 25.0 [3.2 to 65.1]
Statistical Analysis 1: Comparison: Advanced Cutaneous Melanoma; Test type: Superiority; p = 0.0216, Exact Binomial Distribution — One-sided p-value. The ORR was deemed clinically meaningful if the lower bound of the 95% confidence interval exceeded 10% (p<0.0250)

4. Secondary Outcome: ORR Per Investigator Assessment Using RECIST 1.1
Description: The ORR, using RECIST 1.1 criteria, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) at any time during the study, based on Investigator assessment.
Time Frame: Up to 24 months
Population: The FAS population consisted of all allocated participants who had measurable lesions at the Baseline scan as assessed by Investigator review and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
Number analyzed (Participants) | 34 | 8
Percentage of Participants | 29.4 [15.1 to 47.5] | 37.5 [8.5 to 75.5]

5. Secondary Outcome: ORR Per Central Radiology Review Using Immune-related Response Criteria (irRC)
Description: The ORR, using irRC, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (irCR; complete disappearance of all tumor lesions, whether measureable or not, and no new lesions) or a Partial Response (irPR; decrease in sum of the products of the 2 largest perpendicular diameters of 50% or greater) at any time during the study, based on central radiology review.
Time Frame: Up to 24 months
Population: The FAS population consisted of all allocated participants who had irRC measurable lesions at the Baseline scan as assessed by central radiology review and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
Number analyzed (Participants) | 23 | 8
Percentage of Participants | 30.4 [13.2 to 52.9] | 25.0 [3.2 to 65.1]

ADVERSE EVENTS:
Time Frame: All AEs: Up to 30 days after last dose of study drug; Serious AEs: Up to 90 days after last dose of study drug (Up to 27 months)
Description: Safety Population: All participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an adverse event (AE) unless considered related to study drug. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Advanced Cutaneous Melanoma | Advanced Mucosal Melanoma
All-Cause Mortality (participants affected / at risk) | 2/34 | 1/8
Serious Adverse Events (participants affected / at risk) | 13/34 | 4/8
Other Adverse Events (participants affected / at risk) | 34/34 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Cutaneous Melanoma (N=34) | Advanced Mucosal Melanoma (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Death (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Cutaneous Melanoma (N=34) | Advanced Mucosal Melanoma (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 6 (6) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (10) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 5 (7) | 1 (3)
Pyrexia (General disorders) | 8 (13) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 14 (25) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvar erosion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (20) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT02180061/Prot_SAP_000.pdf